CLINICAL TRIAL: NCT05984095
Title: Pelvic Floor Rehabilitation in Females With Multiple Sclerosis: Comparison of Two Telerehabilitation Protocols
Brief Title: Multiple Sclerosis Pelvic Floor Telerehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Trieste (Other)
Responsible Party: Principal Investigator, Alex Buoite Stella, Research fellow, University of Trieste
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Fisioterapia1907
Record Dates: First submitted 2023-08-01; First posted 2023-08-09 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Pelvic Floor; Telerehabilitation; Exercise
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The investigator in charge of reviewing the questionnaires and calculating the scores was not informed about the group of the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SELF (Active Comparator): All the participants in the SELF group were asked to participate in 10 sessions of 45 minutes of pelvic floor training and exercises, once every 5 days. The exercises were available in pre-recorded videos and the participants were allowed to access it when and where they preferred, respecting the requested frequency. No supervision was provided during the trainings.
  Interventions: Other: Telerehabilitation
- REMOTE (Experimental): All the participants in the REMOTE group were asked to participate in 10 sessions of 45 minutes of pelvic floor training and exercises, once every 5 days. The exercises were shown and monitored remotely during a one-to-one videocall with a physiotherapist.
  Interventions: Other: Telerehabilitation

INTERVENTIONS:
Other: Telerehabilitation — The intervention was administered in a telerehabilitation fashion through a videocall on the phone or tablet, by a physiotherapist, in a one-to-one session.

SUMMARY:
The goal of this clinical trial is to compare the effects of two different pelvic floor telerehabilitation protocols on selected measures of quality of life and health in females with relapsing-remitting Multiple Sclerosis (rrMS). The main questions it aims to answer are:

* Is telerehabilitation sufficient to improve quality of life and health in females with rrMS, in particular dedicated to pelvic floor training?
* Are self-administered training protocols or remotely-supervised training protocols equally effective?

Participants will be randomized to two intervention groups: a self-administered training protocol (SELF) and a remotely-supervised (REMOTE) training protocol. Both protocols will consist in 10 sessions of pelvic floor training lasting 45 min each, once every 5 days.

At the start and at the end of the protocol, all participants will complete 6 questionnaires regarding pain, quality of life and health.

DETAILED DESCRIPTION:
In this study, the authors aim to evaluate the efficacy of two telerehabilitation protocols dedicated to pelvic floor and urogynecological health in females with relapsing-remitting Multiple Sclerosis (rrMS).

In particular, the included participants will be randomized to:

* SELF protocol: 10 sessions of pelvic floor exercises, self-administered with a set of videos where a physiotherapist showed the different exercises in order to complete a 45 minutes session.
* REMOTE protocol: 10 sessions of pelvic floor exercises, remotely conducted and supervised by a physiotherapist with a one-to-one videocall, showing and monitoring the exercises in order to complete a 45 minutes session.

One week before the first session and one week after the last session, all the participants will be asked to complete a set of surveys and questionnaires to investigate participants' pain perception, reported quality of life and health-related parameters.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of relapsing remitting Multiple Sclerosis confirmed by a neurologist and based on the McDonald criteria from not less than 1 y
* EDSS <4.5
* self reported symptoms of urinary incontinency

Exclusion Criteria:

* females in menopause
* previous history of bladder or urogynaecological surgery
* previous history of major abdominal surgery
* females with a delivery < 6 months from the start of the study
* BMI > 30

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-25 (Actual)

PRIMARY OUTCOMES:
Pain perception | At baseline (1 week prior the first telerehabilitation session) and after the protocol (1 week after the last telerehabilitation session)
  Quantification of the perceived pain with a numeric rating scale (NRS, score 0-10 where 10 means unbearable plain), and a body chart
Depression symptoms | At baseline (1 week prior the first telerehabilitation session) and after the protocol (1 week after the last telerehabilitation session)
  Evaluation of depression symptoms with the Beck Depression Inventory Scale (BDI, 0-63, higher the score worse the depression)
Perceived quality of life | At baseline (1 week prior the first telerehabilitation session) and after the protocol (1 week after the last telerehabilitation session)
  Evaluation of the perceived quality of life with the Short Form Health Survey 36 (SF-36, 0-100 for each domain, higher the score better the quality of life)
Sexual health | At baseline (1 week prior the first telerehabilitation session) and after the protocol (1 week after the last telerehabilitation session)
  Evaluation of the perceived sexual health with the female sexual function index (FSFI, 1-5 for each item, greater score indicating greater levels of sexual functioning)
Urinary incontinence symptoms | At baseline (1 week prior the first telerehabilitation session) and after the protocol (1 week after the last telerehabilitation session)
  Evaluation of urinary incontinence symptoms with the International Consultation on Incontinence Questionnaire (ICIQ, 0-21, higher the score worse the symptoms)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Manganotti, MD PhD, Study Chair — University of Trieste
Locations (1):
- CdL in Fisioterapia, Trieste, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Deodato M, Fornasaro M, Martini M, Zelesnich F, Sartori A, Galmonte A, Buoite Stella A, Manganotti P. Comparison of different telerehabilitation protocols for urogenital symptoms in females with multiple sclerosis: a randomized controlled trial. Neurol Sci. 2024 Nov;45(11):5501-5509. doi: 10.1007/s10072-024-07742-y. Epub 2024 Sep 3. PMID 39223424